CLINICAL TRIAL: NCT05800379
Title: Study on Hospitalization of Children With Bronchial Asthma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Kunling Shen, professor, Beijing Children's Hospital
Other Study IDs: BCH Lung 010
Record Dates: First submitted 2023-03-01; First posted 2023-04-05 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Asthma in Children
Keywords: asthma; children; mucus plug; Flexible bronchoscope
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bronchial asthma is the most common chronic respiratory disease in children. At present, more attention has been paid to the treatment of airway inflammation and smooth muscle spasm, while the related research on the risk factors of asthma attack, mucus plug formation and its effect on asthma has been ignored. This study was a retrospective study. Children hospitalized for acute exacerbation of asthma from 2016 to 2021 were selected as the research objects. The clinical manifestations, bronchoscopy results and lung CT results of children hospitalized for acute exacerbation of asthma were summarized. To analyze the risk factors of acute exacerbation, clinical characteristics, risk factors of mucus plug formation in hospitalized children with asthma, and the safety and efficacy of flexible bronchoscopy in the diagnosis and treatment of hospitalized children with asthma. The discharged children were investigated by written or online questionnaires to understand the acute attack of asthma, control level, compliance, appliability of the China Children's Asthma Action Plan, family management and medical utilization of children with asthma after discharge.

DETAILED DESCRIPTION:
Asthma is the most common chronic respiratory disease in children. The prevalence of asthma in children in China increased by nearly 50% in 2010 compared with 2000, and the proportion of children hospitalized for asthma exacerbation also increased. China has a large population base, and the number of children with asthma is large. Acute asthma attack is mainly characterized by airway smooth muscle contraction and mucus plug obstruction. At present, more attention has been paid to the treatment of airway mucosal inflammation and smooth muscle spasm, while the related research on the risk factors of asthma acute attack, mucus plug formation and its effect on asthma has been ignored. Bronchoscopy can directly and effectively remove the mucus plug formed in the airway of children with asthma, but there is a lack of clear application standards and procedures. Identifying the risk factors of mucus plug formation in hospitalized children with asthma exacerbation, identifying mucus plug, timely and targeted treatment, and education and training after discharge are of great significance to reduce the hospitalization rate and mortality.This study was a retrospective study. Children hospitalized for acute exacerbation of asthma from 2016 to 2021 were selected as the research objects. The clinical manifestations, bronchoscopy results and lung CT results of children hospitalized for acute exacerbation of asthma were summarized. To analyze the risk factors of acute exacerbation, clinical characteristics, risk factors of mucus plug formation in hospitalized children with asthma, and the safety and efficacy of flexible bronchoscopy in the diagnosis and treatment of hospitalized children with asthma. The discharged children were investigated by written or online questionnaires to understand the acute attack of asthma, control level, compliance, appliability of the China Children's Asthma Action Plan, family management and medical utilization of children with asthma after discharge.

ELIGIBILITY:
Inclusion Criteria:

• Children admitted with acute episodes of asthma between January 2016 and December 2021

Exclusion Criteria:

* Basic information is incomplete
* Lack of relevant information on diagnosis and treatment after admission
* Those who disagree with the telephone follow-up
* Basic diseases such as heart, liver and kidney
* Children with primary or secondary immunodeficiency, genetic metabolic diseases, tumors, or after organ or hematopoietic stem cell transplantation
* Active pulmonary tuberculosis and children with a history of asthma who are hospitalized for other reasons

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children admitted with acute episodes of asthma
Sampling Method: Non-Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics of hospitalized children with acute asthma attack | From January 2016 to December 2021
  clinical characteristics includes: age, sex, asthma severity (mild, severe), asthma inducing factors(infection, allergy, smoke, excerise) and hospitalization expenses
Influencing factors of acute attack severity in hospitalized children with asthma | From January 2016 to December 2021
  age, sex, allergy history, birth history, family history, the severity of asthma exacerbation, lung function and lung computed tomography
Risk factors for acute exacerbation of asthma with respiratory failure in children | From January 2016 to December 2021
  The proportion of children hospitalized for acute exacerbation of asthma with respiratory failure, and age, sex, allergy history（with or without）, family history (asthma, atopic dermatitis,rhinitis and allergy), the severity of asthma exacerbation(mild, severe), lung function (normal, abnormal) and lung computed tomography(normal, abnormal)
Risk factors for mucus plug formation in hospitalized children with asthma exacerbation | From January 2016 to December 2021
  The results of lung CT examination in children with asthma(normal, abnormal), the incidence of mucus plug in hospitalized children with asthma
Identification of mucus plugs in hospitalized children with asthma | From January 2016 to December 2021
  Using mucus scoring system which was based on bronchopulmonary segmental anatomy identified mucus plugs in hospitalized children with asthma. Each bronchopulmonary segment was given a score of 1 (mucus plug present) or 0 (mucus plug absent). The segment scores of each lobe were summed to generate a total mucus score for both lungs, yielding a mucus score ranging from 0-20.

CONTACTS AND LOCATIONS:
Overall Officials: kunling shen, doctor, Principal Investigator — Beijing Children's Hospital
Locations (1):
- Beijing Children's Hospital affiliated to Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han P, Yin J, Zou H, Jiao A, Liu Y, Shen K. Exploring the types of airway inflammation in hospitalized children with asthma. BMC Pediatr. 2025 May 7;25(1):359. doi: 10.1186/s12887-025-05596-7. PMID 40329237